CLINICAL TRIAL: NCT04706923
Title: A Phase IIa, Open-label, Multiple Ascending Dose Confirmation Study of the Safety and Tolerability of Intravenous Administration of Brincidofovir in Subjects With Adenovirus Infection or Cytomegalovirus Infection
Brief Title: A Phase 2a Study of IV BCV in Subjects With Adenovirus Infection
Acronym: ATHENA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCV-PA01
Record Dates: First submitted 2021-01-05; First posted 2021-01-13 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Adenovirus Infections; Cytomegalovirus Infection
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BCV 0.2mg/kg BIW (Experimental): BCV: 0.2 mg/kg administered as a continuous IV infusion over 2 hours
  Interventions: Drug: BCV
- BCV 0.3mg/kg BIW (Experimental): BCV: 0.3 mg/kg administered as a continuous IV infusion over 2 hours
  Interventions: Drug: BCV
- BCV 0.4 mg/kg BIW (Experimental): BCV: 0.4 mg/kg administered as a continuous IV infusion over 2 hours
  Interventions: Drug: BCV
- BCV 0.4 mg/kg QW (Experimental): BCV: 0.4 mg/kg administered as a continuous IV infusion over 2 hours
  Interventions: Drug: BCV

INTERVENTIONS:
Drug: BCV — Brincidofovir (BCV) is a lipid conjugate of the antiviral cidofovir that enables optimal intracellular levels of the active drug.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of intravenous (IV) brincidofovir (BCV; SyB V-1901) 0.2 mg/kg, 0.3 mg/kg or 0.4 mg/kg dosed twice weekly (BIW) or 0.4 mg/kg dosed once weekly (QW) for 4 weeks in subjects with AdV, and IV BCV in subjects with CMV

DETAILED DESCRIPTION:
This is a Phase IIa, open-label, multiple ascending dose confirmation, multicenter study to evaluate the safety and tolerability of intravenous Brincidofovir (BCV, SyB V-1901) 0.2 mg/kg, 0.3 mg/kg, or 0.4 mg/kg dosed BIW or 0.4 mg/kg dosed QW (Cohorts 1 to 4) in adult and pediatric subjects with AdV viremia, and IV BCV in subjects with CMV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 2 months and older at the time of informed consent.
* AdV DNA viremia >10,000 copies/mL from a single sample, or 2 samples greater than 48 hours apart with the second result higher than the first and both greater than 1000 copies/mL, from the data obtained from the designated central virology laboratory of the local laboratory using the blood sample(s) collected informed consent has been obtained and within 7 days prior to Day 1 (AdV DNA viremia results collected within the 7 day window, but prior to consent may be used if the Informed Consent Form (ICF) signed by the subject provides approval) . CMV viremia with or without evidence of tissue invasive CMV disease. For laboratory results that are generated in units other than copies/mL or IU/mL, please refer to the testing laboratory for guidance on the appropriate conversion calculation.
* Either (a) have disseminated AdV disease or (b) have an underlying immunocompromised state, and have asymptomatic AdV infection or localized AdV disease.
* In the judgment of the investigator, be in a serious condition to be treated with intravenous cidofovir for AdV.

Exclusion Criteria:

* Subjects who weigh ≥120 kg.
* NIH/NCI CTCAE (United States [US] National Institutes of Health [NIH]/National Cancer Institute) Grade 2 or higher diarrhea (i.e., increase of ≥ 4 stools per day over usual pre-transplant stool output) within 7 days prior to Day 1.
* NIH Stage 4 acute GVHD of the skin (i.e., generalized erythroderma with bullous formation) within 7 days prior to Day 1.
* NIH Stage 2 or higher acute GVHD of the liver function (i.e., bilirubin >3 mg/dL [SI: >51 μmol/L]) within 7 days prior to Day 1.
* NIH Stage 2 or higher acute GVHD of the gut (i.e., diarrhea >556 mL/m2/day for pediatric subjects [or >1000 mL/day for young adults as applicable, at centers in the United States only], or severe abdominal pain with or without ileus) within 7 days prior to Day 1.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety will be evaluated based on incidence and severity of Adverse Events, Serious Adverse Events and laboratory assessments. | From initiation of BCV administration up to 19 weeks
  Safety will be evaluated based on incidence and severity of Adverse Events, Serious Adverse Events and laboratory assessments.
Antiviral Effects | From initiation of BCV administration up to 9 weeks
  Change from baseline AdV viremia in plasma measured on Day 1 and weekly throughout the study.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Research Site, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.symbiopharma.com/en/pipeline/overview.html